CLINICAL TRIAL: NCT07314970
Title: Impact of the Practitioner's Discourse on the Mother's Decision Regarding the Mode of Delivery in Cases of Breech Presentation
Brief Title: Discourse on the Mother's Decision Regarding the Mode of Delivery in Cases of Breech Presentation
Acronym: DISCOURS-SIEGE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9537
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Breech Presentation
Keywords: Breech Presentation
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Doctor with a primary focus on Obstetrics: * Practicing in a University Hospital in the Grand Est region (Besançon, Reims, Strasbourg, Nancy)
  * Agreeing to complete the self-administered questionnaire anonymously.
  Interventions: Other: To complete a questionnaire
- Adult woman (≥ 18 years old): * Gave birth in 2024 at a university hospital in the Grand Est region (Besançon, Reims, Strasbourg, Nancy)
  * Breech delivery > 37 weeks gestation
  * Agree to complete the self-administered questionnaire anonymously.
  Interventions: Other: To complete a questionnaire

INTERVENTIONS:
Other: To complete a questionnaire — Doctor and Adult woman agreeing to complete the self-administered questionnaire anonymously.

SUMMARY:
Breech presentation is a common occurrence in routine practice, occurring in 3-4% of all term pregnancies. Despite its frequency, breech presentation at term remains a subject of considerable controversy within the medical community. This results in differing management approaches depending on the country, the center, and the practitioner. Indeed, from a pathophysiological perspective, during a breech delivery, the fetal head is the last segment to descend into the maternal pelvis. This is the largest fetal segment in terms of volume. Furthermore, the fetal head cannot accommodate itself to the maternal pelvis through plastic deformation. This presentation can therefore lead to specific complications that may be life-threatening for the unborn child.

Despite its frequency, breech presentation at term remains a subject of considerable controversy within the medical community regarding the management of labor. In the 2000s, a randomized trial called the TERM BREECH TRIAL found a neonatal benefit of planned cesarean section compared to vaginal delivery of a breech fetus (prevention of perinatal death in 1% of cases). This resulted in a significant increase in the rate of planned cesarean sections for breech presentation worldwide. However, numerous more recent studies (notably PREMODA in France) have highlighted the many biases of the Term Breech Trial, and various literature reviews (including the 2015 Cochrane review) have demonstrated lower perinatal morbidity than that found by Hannah's team. In 2020, the CNGOF (National College of Gynecologists and Obstetricians of France) published new recommendations on the management of breech presentations at the end of pregnancy, proposing vaginal delivery as a possible alternative to a planned cesarean section, provided that the patient receives clear and honest information (benefits and risks of each delivery method). The choice of delivery method must be made in consultation with the patient after a dedicated consultation. Since these recommendations were published, management practices still vary between hospitals despite fairly precise guidelines.

ELIGIBILITY:
Inclusion Criteria:

Regarding practitioners:

* Doctor with a medical degree (Junior Doctor, Clinical Assistant, Hospital Practitioner, University Professor of Obstetrics), with a primary focus on Obstetrics
* Practicing in a University Hospital in the Grand Est region (Besançon, Reims, Strasbourg, Nancy)
* Agreeing to complete the self-administered questionnaire anonymously.

Regarding patients:

* Patient of legal age (≥ 18 years)
* Having given birth in 2024 in a university hospital in the Grand-Est region (Besançon, Reims, Strasbourg, Nancy)
* Delivery of a breech fetus > 37 weeks of gestation
* Agreeing to answer the self-administered questionnaire anonymously.

Exclusion Criteria:

Regarding practitioners:

Other primary activity than obstetrics

Regarding patients:

* Minor patient at the time of delivery
* Patient who had a cesarean section due to a uterine scar and maternal desire.
* Patients with a history of uterine scarring or the presence of obstruction previa were also excluded due to the impossibility of authorizing vaginal delivery, regardless of fetal presentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Doctor with a medical degree (Junior Doctor, Clinical Assistant, Hospital Practitioner, University Professor of Obstetrics), with a primary focus on Obstetrics.
  * Patient of legal age (≥ 18 years)
  * Having given birth in 2024 in a university hospital in the Grand-Est region (Besançon, Reims, Strasbourg, Nancy)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Overall satisfaction of women who gave birth to a breech fetus regarding their medical care | Up to 12 months
  Questionnaire from the book "The Joyful and Relaxed Pregnancy Guide"
  Score from 0 to 10:
  0 = Not at all satisfied 5 = Partially satisfied 10 = Completely satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologique et d'Obstétrique - CHU de Strasbourg - France, Strasbourg, France